CLINICAL TRIAL: NCT05768152
Title: Repeated Low-level Red-light Therapy in High Myopia Children and Teenagers: a Prospective Single-arm Study
Brief Title: Repeated Low-Level Red-Light Therapy Shortens Axial Length
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second People's Hospital of Foshan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: (2022)-0131
Record Dates: First submitted 2023-02-20; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: High Myopia; Axial Length; Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Repeated low-level red-light (RLRL) therapy (Experimental): single vision spectacles & RLRL
  Interventions: Device: RLRL

INTERVENTIONS:
Device: RLRL — RLRL will be performed twice per day with an interval of at least 4 hours, each treatment last 3 minutes, in addition to single vision spectacles with power for correcting distance refraction.

SUMMARY:
The purpose of this clinical trial is to investigate the incidence and magnitude of axial length shortening after repeated low-level red-light therapy in high myopia children and teenagers.

DETAILED DESCRIPTION:
High myopia has become a major public concern globally, which is characterized by excessive axial elongation of the eyeball. Axial elongation is accompanied by mechanical stretching and thinning of the choroid and sclera, causing vision-threatening complications. Repeated low-level red-light (RLRL) therapy is an emerging effective and safe therapy for myopia control. Previous clinical trials in China have observed clinically significant axial shortening after RLRL treatment.

The purpose of this study is to investigate and identify possible mechanism for axial length (AL) shortening after 12-month RLRL therapy in highly myopic children and teenagers aged 8-18 years. In addition to single vision spectacles, subjects will receive RLRL treatment at home under supervision of the parents/guardians according to a standard protocol. Axial length, visual acuity, cycloplegic spherical equivalent refraction, slit lamp, fundus camera and optical coherence tomography/angiography will be measured at 1-, 3-, 6- and 12-month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of consent.
2. Age: ≥ 8 and ≤ 18 years at enrolment.
3. High myopia: cycloplegic sphere of -6.00 diopters (D) or greater in both eyes.
4. Willing and able to participate in all required activities of the study.
5. The children currently on myopia control treatment can be recruited if myopia control treatments (including but not limited to atropine, orthokeratology, rigid gas-permeable lenses, defocus spectacles, etc.) are discontinued for at least 2 weeks.
6. Normal fundus, tessellated fundus or with peripapillary diffuse chorioretinal atrophy.

Exclusion Criteria:

1. Secondary myopia, such as a history of retinopathy of prematurity or neonatal problems, or syndromic myopia with a known genetic disease or connective tissue disorders, such as Stickler or Marfan syndrome.
2. Pathologic myopia with signs of macula-involving diffuse chorioretinal atrophy, patchy chorioretinal atrophy, macular atrophy, lacquer cracks, myopic choroidal neovascularization or Fuchs' spots.
3. Strabismus and binocular vision abnormalities in either eye.
4. Previous any intraocular surgery affecting refractive status.
5. Other reasons, including but not limited to ocular or other systemic abnormalities, that the physician may consider inappropriate for enrolment.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of axial length shortening greater than 0.05 mm | 12 months
  Incidence rate of axial length shortening > 0.05 mm is characterized as the ratio of the number of participants whose axial length has shortened by greater than 0.05 mm to the total number of participants. Axial length (mm) is measured using the IOL Master.

SECONDARY OUTCOMES:
Incidence rates of axial length reduction greater than 0.10 mm and 0.20 mm | 12 months
  Incidence rates of axial length shortening > 0.10 mm and 0.20 mm are characterized as the ratio of the number of participants whose axial length has shortened by greater than 0.10 mm and 0.20 mm to the total number of participants. Axial length (mm) is measured using the IOL Master.
Magnitude of axial length shortening among shortened eyes | 12 months
  The magnitude of axial length shortening is characterized as the amount of axial length reduction in eyes with axial shortening. Axial length (mm) is measured using the IOL Master.
Changes in choroidal thickness (μm) | 1, 3, 6 and 12 months
  Changes in choroidal thickness are characterized as the difference between each follow-up visit and corresponding baseline values which are measured using the optical coherence tomography.
Changes in axial length (mm) | 1, 3, 6 and 12 months
  Changes of axial length is characterized as the difference between each follow-up visit and baseline values which are measured using the IOL Master.
Changes in corneal curvature (mm) | 1, 3, 6 and 12 months
  Changes of corneal curvature is characterized as the difference between each follow-up visit and baseline values which are measured using the IOL Master.
Changes in anterior chamber depth (mm) | 1, 3, 6 and 12 months
  Changes of anterior chamber depth is characterized as the difference between each follow-up visit and baseline values which are measured using the IOL Master.
Changes in white to white (mm) | 1, 3, 6 and 12 months
  Changes of white to white is characterized as the difference between each follow-up visit and baseline values which are measured using the IOL Master.
Change of cycloplegic spherical equivalent refraction | 1, 3, 6 and 12 months
  Cycloplegic spherical equivalent change (Diopter, D) is characterized as the difference between each follow-up visit and baseline values. Refraction with full cycloplegia is performed with an autorefractor. The data on spherical and cylindrical power and axis is automatically extracted from the autorefractor. The spherical equivalent power (D) is calculated as the spherical power (D) plus half of the cylindrical power (D).
Change of pathologic myopia fundus META-PM grading | 1, 3, 6 and 12 months
  The fundus images are classified based on META-PM classification system. Color fundus images are obtained using the fundus camera.
Change in best corrected visual acuity | 1, 3, 6 and 12 months
  Best corrected visual acuity change is characterized as the difference between each follow-up visit and baseline values. Visual acuity is assessed using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart with standard illumination at a distance of 4 meters.
Incidence of self-reported adverse events | 1, 3, 6 and 12 months
  Incidence of self-reported adverse events is the rate of self-reported adverse events over a specified period for all the subjects. Subjects are asked to report any treatment-emergent adverse events, including but not limited to glare, flash blindness, and afterimages.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second People's Hospital of Foshan, Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared as open data after proper anonymization.